CLINICAL TRIAL: NCT03428360
Title: An Open-Label, Safety and Tolerability Study of Chronic Intermittent Use of Diazepam Buccal Film (DBF) in Pediatric, Adolescent and Adult Subjects With Epilepsy
Brief Title: Safety and Tolerability Study of Diazepam Buccal Film (DBF) in Subjects With Epilepsy
Acronym: DBF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aquestive Therapeutics (Industry)
Collaborators: Syneos Health (Other); Covance (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 42-1703
Record Dates: First submitted 2017-12-18; First posted 2018-02-09 (Actual); Results first posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Epilepsy
Keywords: Seizure
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Intervention Model Description: The study population was male or female pediatric, adolescent, and adult subjects with a clinical diagnosis of epilepsy and with bouts of increased seizure activity, frequent breakthrough seizures, seizure clusters, or cluster seizures and who were on chronic, intermittent use of rescue medication (eg, Diastat AcuDial or other benzodiazepine).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Subjects with Epilepsy (Experimental): Male or female subjects between the ages of 2 and 65 years who had an established diagnosis of epilepsy exhibited by motor seizures with clear alteration of awareness, and while on a regimen of anti-epileptic medication(s), still experienced bouts of seizures (frequent breakthrough seizures, eg, seizure clusters) and who, in the opinion of the Investigator, could need benzodiazepine intervention for seizure control at least 1 time a month on average. Subjects must have been on at least 1 concomitant anti-epileptic drug at screening.
  Interventions: Drug: Diazepam Buccal Soluble Film 5, 7.5,10, 12.5,15 or 17.5 mg with individual dose determined according to age and weight category

INTERVENTIONS:
Drug: Diazepam Buccal Soluble Film 5, 7.5,10, 12.5,15 or 17.5 mg with individual dose determined according to age and weight category — The subjects in this study administered DBF themselves or with the help of a caregiver, (trained by the study site staff in study drug administration and documentation) in the same setting as they typically used the diazepam rectal gel or other rescue medication, without the presence of study staff.
  Other Names: DBF, Diazepam Buccal Film (Aquestive Therapeutics)

SUMMARY:
This Phase 3, multicenter, open-label study of chronic, intermittent use of study drug (DBF) is designed to evaluate the safety and tolerability of the buccal formulation of diazepam in children, adolescents and adults with intermittent, stereotypic episodes of frequent seizure activity (eg, seizure clusters) that are distinct from the subject's usual seizure pattern.

DETAILED DESCRIPTION:
The Primary objective of the study is to assess the safety and tolerability of DBF (study drug) administered a minimum of 3 times to subjects with epilepsy for the treatment of seizures over a minimum 6-month period.

Secondary objectives:

* To evaluate the usability of study drug as assessed by the ability of caregivers/subjects to administer study drug based on the Instructions for Use (IFU).
* To evaluate the Quality of Life (QoL) of the subjects during the study drug treatment period as assessed by use of age-appropriate epilepsy scales over a minimum 6-month period.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male subject between the ages of 2 and 65 years of age, inclusive
2. Written informed consent to participate in the study
3. Subject has an established diagnosis of epilepsy either partial or generalized epilepsy with motor seizures with clear alteration of awareness, and while on a regimen of anti-epileptic medication(s), still experiences bouts of seizures (frequent break through seizures, e.g. Acute Repetitive Seizures (ARS) or seizure clusters) and who, in the opinion of the Investigator, may need benzodiazepine intervention for seizure control at least 1 time a month on average.
4. Caregiver, if needed for subject, provides written informed consent and is able to administer study drug in the event of a seizure.
5. Female subjects ≥12 years of age have a negative serum pregnancy test at screening. Female subjects of childbearing potential, (not surgically sterile or less than 2 years postmenopausal), must have a partner who is sterile, agrees to abstinence, be practicing double barrier contraception or using an FDA approved contraceptive (e.g., licensed hormonal or barrier methods) for greater than 2 months prior to screening visit and commit to an acceptable form of birth control for the duration of the study and for 30 days after the study
6. No aspects of the medical history and/or the physical-neurological examination that at the judgment of the Investigator, in consultation with the Sponsor, will interfere with administration or absorption of study drug, or could evolve into a safety issue
7. No clinically significant abnormal findings on the electrocardiogram (QTcF≤450 msec for males and QTcF≤470 msec for females)
8. Subject and caregiver must be willing to comply with all study visits and all required study procedures

Exclusion Criteria:

1. A history of clinically significant gastrointestinal, renal/genitourinary, hepatic, hematologic, dermatologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease, or any other clinically significant abnormalities, such as physical examination, vital signs, laboratory tests or ECG at Screening or Baseline which in the opinion of the investigator require further investigation or treatment or which may interfere with study procedures or safety or other medical conditions (e.g., cardiac, respiratory, gastrointestinal, psychiatric, renal disease) which are not adequately and stably controlled, or which in the opinion of the investigator(s) could affect the subject's safety or interfere with the study assessments or any other condition which, in the opinion of the Investigator, would jeopardize the safety of the subject
2. Subject has had significant traumatic injury, major surgery or open biopsy within 30 days prior to study screening
3. Subject with an active major depression or a past suicide attempt, or any suicidal ideation of 4, or 5 or any suicidal behavior in lifetime using Columbia-Suicide Severity Rating Scale(C-SSRS). The pediatric C-SSRS should be used for subjects 6 to 11 years of age. The adult C-SSRS should be used for subjects ≥12 years of age. Note that this exclusion is only applicable to cognitive-appropriate subjects who are able to understand and complete the Suicide Rating Scale
4. A history of allergic or adverse responses to diazepam or any other benzodiazepine
5. Participation in a clinical trial other than MonoSol Rx Phase 2 studies 160325 and 160326 within 30 days prior to Day 0. Participation in an observational (non-interventional) study is not an exclusion, provided that there are no scheduling conflicts with this study. Received any other investigational medication (unless it can be documented that the subject received only placebo) or device within 8 weeks or 5 half-lives (whichever is longer) before assignment to study drug treatment
6. Lactating female or positive serum pregnancy test (ß-hCG) at screening for female subjects ≥12 years of age
7. Positive blood screen for HIV, HbSAg, or Hepatitis C, or a positive urine screen for alcohol or drugs of abuse, except marijuana use for medicinal indications. When marijuana is or was used for medicinal indications in the opinion of the Investigator, it is not considered as drug abuse and the subject can be enrolled in states where medical marijuana use is legal, even if the marijuana metabolites in the urine revealed as positive

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Slatko, Study Director — Aquestive Therapeutics
Locations (6):
- United States (6):
  - Hawaii Neuroscience Center, Honolulu, Hawaii
  - Consultants in Epilepsy and Neurology, PLLC, Boise, Idaho
  - Clinical Research Center of New Jersey (CRCNJ), Voorhees Township, New Jersey
  - OnSite Clinical Solutions LLC, Charlotte, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Austin Epilepsy Care Center, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 150 subjects with epilepsy passed screening but 1 was never enrolled
Pre-assignment Details: 149 were enrolled but only 130 received at least 1 dose of study drug and were included in the analyses
Groups:
- Safety Set: Male or female subjects between the ages of 2 and 65 years who had an established diagnosis of epilepsy exhibited by motor seizures with clear alteration of awareness, and while on a regimen of anti-epileptic medication(s), still experienced bouts of seizures (frequent breakthrough seizures, eg, seizure clusters) and who, in the opinion of the Investigator, could need benzodiazepine intervention for seizure control at least 1 time a month on average. Subjects must have been on at least 1 concomitant anti-epileptic drug at screening.
  Diazepam Buccal Soluble Film 5, 7.5,10, 12.5,15 or 17.5 mg with individual dose determined according to age and weight category: The subjects administered DBF themselves or with the help of a caregiver, (trained by the study site staff in study drug administration and documentation) in the same setting as they typically used the diazepam rectal gel or other rescue medication, without the presence of study staff.
Period: Overall Study
Arm/Group | Safety Set
Started | 130
Completed | 90
Not Completed | 40
Not completed — Informed consent withdrawn | 5
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 5
Not completed — Physician Decision | 2
Not completed — Informed consent withdrawn | 5
Not completed — Study terminated by sponsor | 10
Not completed — Non-compliant with study | 1
Not completed — Non-compliant with study drug | 3
Not completed — Death | 3
Not completed — Adverse Event | 1
Not completed — Not on antiepileptic drug | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: Enrolled subjects with epilepsy who received at least 1 dose of study drug
Groups:
- Safety Analysis Set: Enrolled Subjects With Epilepsy Who Received at Least 1 Dose of Study Drug: Male or female subjects between the ages of 2 and 65 years who had an established diagnosis of epilepsy exhibited by motor seizures with clear alteration of awareness, and while on a regimen of anti-epileptic medication(s), still experienced bouts of seizures (frequent breakthrough seizures, eg, seizure clusters) and who, in the opinion of the Investigator, could need benzodiazepine intervention for seizure control at least 1 time a month on average. Subjects must have been on at least 1 concomitant anti-epileptic drug at screening.
  Diazepam Buccal Soluble Film 5, 7.5,10, 12.5,15 or 17.5 mg with individual dose determined according to age and weight category: The subjects in this study administered DBF themselves or with the help of a caregiver, (trained by the study site staff in study drug administration and documentation) in the same setting as they typically used the diazepam rectal gel or other rescue medication, without the presence of study staff.
Arm/Group | Safety Analysis Set: Enrolled Subjects With Epilepsy Who Received at Least 1 Dose of Study Drug
Number analyzed (Participants) | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.9 (13.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29
  Not Hispanic or Latino | 99
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 6
  Black or African American | 12
  White | 99
  More than one race | 8
  Unknown or Not Reported | 0
Body Mass Index (kg/m^2 [Mean (Standard Deviation); unit: kg/m^2] | 24.108 (6.8148)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects in the Safety Analysis Set With at Least 1 Treatment-emergent Adverse Event (TEAE)
Description: A TEAE was defined as any adverse event with onset date on the day of or after administration of study drug including relationship and severity.
Time Frame: Adverse events (AEs) were recorded from Day 1 through the last study contact (Month 7 telephone contact).
Population: Subjects who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Analysis Set: Enrolled Subjects With Epilepsy Who Received at Least 1 Dose of Study Drug
Number analyzed (Participants) | 130
Participants
  At least 1 TEAE | 84
  At least 1 severe TEAE | 14
  At least 1 study drug related TEAE | 10
  At least 1 severe and related TEAE | 1
  At least 1 serious TEAE | 18
  At least 1 serious and related TEAE | 1

2. Primary Outcome: Number of Subjects in Safety Analysis Set With Adverse Events of Special Interest (AESI)
Description: A.Oral irritation related AEs including but not limited to: buccal mucosal swelling, mouth ulceration, injuries to oral cavity (such as tongue or mucosal laceration, broken tooth, bleeding), erythema, stomatitis, gingivitis, xerostomia, staining, dysphagia, dysgeusia, burning, stinging, tingling.
  B. Abuse related AEs including euphoria, euphoric mood, feeling of relaxation, anger, dissociative effects, hallucinations, psychosis, changes in mood, impaired cognition, attention, psychomotor effects, inappropriate affect, overdose, and misuse.
  C. Other: Respiratory disorders, nervous system disorders
Time Frame: AESIs were recorded from Day 1 through the last study contact (Month 7 telephone contact).
Population: Subjects who received at least 1 dose of study drug
Measure: Number; unit: participants
Arm/Group | Subjects With Epilepsy
Number analyzed (Participants) | 130
participants
  Any adverse event of special interest | 32
  Any oral irritation adverse event | 3
  Any oral safety adverse event | 8
  Any potential abuse related adverse event | 21
  Any abuse related adverse event | 1
  Any other adverse event of special interest | 8

3. Secondary Outcome: Usability Assessment: Number of Use Occasions Where Difficulty in Opening the Outer Packaging Was Recorded.
Description: For each use occasion the following question was asked: Did you have difficulty in opening the outer plastic packaging on this use occasion? Yes
Time Frame: Recorded in an electronic diary after each use of study drug, throughout the course of the study; approximately 6 months
Population: Subjects who received at least 1 dose of study drug (Safety Analysis Set)
Measure: Number; unit: total number of use occasions
Units Other Than Participants: total number of use occasions
Groups:
- Total Use Occasions: Analysis is based upon the total number times the study drug was used over the course of the study - subjects could have multiple use occasions during the study: Total number of use occasions reported was 1348 for the total 130 subjects in the Safety Population
Arm/Group | Total Use Occasions
Number analyzed (Participants) | 130
Number analyzed (total number of use occasions) | 1348
total number of use occasions | 211

4. Secondary Outcome: Usability Assessment: Ability to Open Foil Pouch on Each Use Occasion
Description: For each use occasion the following question was asked: Did you have difficulty in opening the foil pouch on this use occasion? Yes or No
Time Frame: as for outcome 3
Population: Number of subjects reporting use occasions
Measure: Count of Units; unit: total number of use occasions
Units Other Than Participants: total number of use occasions
Groups:
- Study Drug Use Occasions: Total number of use occasions reported over the course of the study; each subject could report multiple use occasions during the study
Arm/Group | Study Drug Use Occasions
Number analyzed (Participants) | 130
Number analyzed (total number of use occasions) | 1348
total number of use occasions
  Yes, I had difficulty opening the foil pouch | 391
  No, I did not have difficulty opening the foil pouch | 957

5. Secondary Outcome: Usability Assessment: Ability to Remove Study Drug From Foil Pouch on Each Use Occasion
Description: For each use occasion the following question was asked: Did you have difficulty in removing study drug from foil pouch on this occasion? Yes or No
Time Frame: as for outcome 3
Population: Subjects who received at least 1 dose of study drug (Safety Analysis Set)
Measure: Count of Units; unit: total number of use occasions rpoeted
Units Other Than Participants: total number of use occasions rpoeted
Groups:
- Study Drug Use Occasions: Total number of use occasions reported during the study; each subject could report multiple use occasions over the course of the study
Arm/Group | Study Drug Use Occasions
Number analyzed (Participants) | 130
Number analyzed (total number of use occasions rpoeted) | 1348
total number of use occasions rpoeted
  Yes, I had difficulty removing study drug from pouch on this occasion | 47
  No, I did not have difficulty removing study drug from the pouch on this occasion | 1301

6. Secondary Outcome: Number of Occasions With Successful Insertion/Retention in Cheek
Description: Of the total number of use occasions over the course of the study, the number of use occasions that were successfully inserted/retained in the cheek
Time Frame: as for outcome 3
Population: Subjects who received at least 1 dose of study drug (Safety Analysis Set)
Measure: Number; unit: Number of events
Units Other Than Participants: total number of use occasions
Arm/Group | Study Drug Use Occasions
Number analyzed (Participants) | 130
Number analyzed (total number of use occasions) | 1348
Number of events | 1330

7. Secondary Outcome: Usability Assessment: Difficulty Inserting DBF Against the Buccal Mucosa (Number of Attempts to Insert Film for Each Use Occasion)
Description: Number of occasions where it took 1 attempt to insert film, Number of occasions where it took 2 attempts to insert film, Number of occasions where it took 3 attempts to insert film, Number of occasions where it took >3 attempts to insert film
Time Frame: as for outcome 3
Population: Subjects who received at least 1 dose of study drug (Safety Analysis Set)
Measure: Number; unit: Number of events
Units Other Than Participants: total number of use occasions
Arm/Group | Study Drug Use Occasions
Number analyzed (Participants) | 130
Number analyzed (total number of use occasions) | 1348
Number of events
  Number of occasions where it required 1 attempt to insert film | 1268
  Number of occasions that required 2 attempts to insert film | 38
  Number of occasions that required 3 attempts to insert film | 18
  Number of occasions that required >3 attempts to insert film | 6

8. Secondary Outcome: Usability Assessment: Number of Occasions Where DBF Was Not Placed or Retained on the Inner Cheek Until Dissolution
Description: Number of occasions where the study drug was not successfully placed and or retained in cheek until the film fully dissolved.
Time Frame: as for outcome 3
Population: Subjects who received at least 1 dose of study drug (Safety Analysis Set)
Measure: Count of Units; unit: total number of use occasions
Units Other Than Participants: total number of use occasions
Arm/Group | Study Drug Use Occasions
Number analyzed (Participants) | 130
Number analyzed (total number of use occasions) | 1348
total number of use occasions | 16

9. Secondary Outcome: Usability Assessment: Reasons for Multiple Placement/Insertion Attempts During a Use Occasion
Description: Reasons for multiple attempts at insertion Multiple choice answer was: Excessive drooling, Clenching jaw / Won't open mouth, Spit out before sticking, Other/None of the above
Time Frame: as for outcome 3
Population: Subjects who received at least 1 dose of study drug (Safety Analysis Set)
Measure: Number; unit: total number of use occasions
Units Other Than Participants: total number of use occasions
Arm/Group | Study Drug Use Occasions
Number analyzed (Participants) | 130
Number analyzed (total number of use occasions) | 1348
total number of use occasions
  Clenching jaw / won't open mouth | 21
  Excessive drooling | 24
  Spit out before sticking | 17
  Other (none of the above) | 33

ADVERSE EVENTS:
Time Frame: Adverse events that started after the first intake of DBF through the Final Visit were considered treatment-emergent adverse events (TEAEs).
Groups:
- Safety Analysis Set: Male or female subjects between the ages of 2 and 65 years who had an established diagnosis of epilepsy exhibited by motor seizures with clear alteration of awareness, and while on a regimen of anti-epileptic medication(s), still experienced bouts of seizures (frequent breakthrough seizures, eg, seizure clusters) and who, in the opinion of the Investigator, could need benzodiazepine intervention for seizure control at least 1 time a month on average. Subjects must have been on at least 1 concomitant anti-epileptic drug at screening.
  Diazepam Buccal Soluble Film 5, 7.5,10, 12.5,15 or 17.5 mg with individual dose determined according to age and weight category: The subjects in this study administered DBF themselves or with the help of a caregiver, (trained by the study site staff in study drug administration and documentation) in the same setting as they typically used the diazepam rectal gel or other rescue medication, without the presence of study staff.
Arm/Group | Safety Analysis Set
All-Cause Mortality (participants affected / at risk) | 3/130
Serious Adverse Events (participants affected / at risk) | 17/130
Other Adverse Events (participants affected / at risk) | 84/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Analysis Set (N=130)
Seizure (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Partial seizure (Nervous system disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Death (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Analysis Set (N=130)
Seizure (Nervous system disorders) | 26 (98)
Somnolence (Nervous system disorders) | 6 (6)
Lethargy (Nervous system disorders) | 4 (5)
Dizziness (Nervous system disorders) | 4 (4)
Headache (Nervous system disorders) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 8 (8)
Sinusitis (Infections and infestations) | 6 (6)
Ear infection (Infections and infestations) | 4 (4)
Vomiting (Gastrointestinal disorders) | 7 (8)
Nausea (Gastrointestinal disorders) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 4 (6)
Fall (Injury, poisoning and procedural complications) | 5 (7)
Skin abrasion (Injury, poisoning and procedural complications) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pyrexia (General disorders) | 7 (12)
Weight decreased (Investigations) | 4 (6)
Weight increased (Investigations) | 4 (6)

LIMITATIONS AND CAVEATS:
Only those subjects who received at least one dose of DBF (130 out of 149) for a breakthrough seizure were included in the Safety Analysis Set.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/60/NCT03428360/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/60/NCT03428360/SAP_001.pdf